CLINICAL TRIAL: NCT04088019
Title: Proportion of Clinical Improvement and Score Comparison of Type 1 Interferon, Transcriptomic Analysis in Idiopathic Uveitis Patients With IGRA Positive Before and After Anti-Tuberculosis Drugs Treatment: Cohort Prospective Study
Brief Title: Proportion of Clinical Improvement & Type 1 Interferon (IFN) Score Changes in Idiopathic Uveitis Patients With Interferon Gamma Release Assay (IGRA) Positive
Status: Recruiting | Type: Observational
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rina, Lecturer, Fakultas Kedokteran Universitas Indonesia
Other Study IDs: 19-06-0769
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis; Uveitis (Manifestation); Anti-Tuberculous Drug Reaction; Tuberculous Uveitis
Keywords: Idiopathic uveitis; IGRA positive; Type 1 interferon; Transcriptomic analysis; Anti-Tuberculosis Therapy
MeSH Terms: conditions — Tuberculosis; Uveitis | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood from the patients are collected in PAXgene blood RNA tubes (QIAGEN). The RNA from the whole blood is extracted and proceed for further examinations (type 1 interferon expression and transcriptomic analysis).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort group: Subjects: idiopathic uveitis with IGRA positive.
  Examinations:
  * Clinical improvement examinations at day 0, second week, week 8, month 3, month 6 and month 12.
  * Blood sampling at day 0, second week, month 6 for analysing type 1 IFN gene expression scoring using RT-qPCR methods.
  Interventions: Drug: Fixed drug combination (FDC) of ATT and Oral steroid

INTERVENTIONS:
Drug: Fixed drug combination (FDC) of ATT and Oral steroid — In the first two week, patients receive FDC of ATT only. Oral steroid start to be given in week three.
  The ATT regiment is continued for up to 6 months or more, in accordance with WHO guidelines. In the first two months the antibiotic combination given consisted of isoniazid (INH), rifampicin, pyrazinamide, and ethambutol. The next four months or continuation phases, the ATT given is rifampicin and isoniazid.
  The following dosage and administration of oral steroids will be given to patients, according to guidelines from the American Journal of Ophthalmologists (Douglas A. Jabs et al, 2000):
  Initial dose: 1mg/kg/day, with maximum adult oral dose 60-80 mg/kg and maintenance dose less than or equal to 10 mg/day. The tapering schedule: Over 40 mg/day, decrease by 10 mg/day every 1-2 weeks, 40-20 mg/day, decrease by 5 mg/day every 1-2 weeks, 20-10 mg/day, decrease by 2.5 mg/day every 1-2 weeks, 10-0 mg/day, decrease by 1 to 2.5 mg/day every 1-4 weeks.

SUMMARY:
The aim of this study is to determine the proportion of clinical improvement, the score changing of type 1 interferon selected gene expression, and analysis of transcriptomics profiling in patients with idiopathic uveitis positive IGRA before and after receiving Anti-Tuberculosis Therapy (ATT).

Hopefully, by conducting this research, we are able to provide valid data that demonstrate the advantages/disadvantages usage of Anti-Tuberculosis Therapy in patients with idiopathic uveitis IGRA positive that correlate with type I IFN. This research is a part of our efforts in discovering bio-marker candidates of idiopathic uveitis IGRA positive clinical patients who will benefit from the ATT administration.

DETAILED DESCRIPTION:
Diagnostic of Idiopathic Uveitis IGRA Positive patients were still unclear. This situation happens because it is still can't be explained if the uveitis from the patients was caused by mycobacterium tuberculosis or not which leads to doubtfulness for Anti-Tuberculosis Treatment (ATT). This study aims to help to provide evidence on whether ATT usage for Idiopathic Uveitis IGRA Positive would bring beneficial impact for the patients. This study will try to analyze the data from clinical improvements, Type 1 Interferon changes, and transcriptomics analysis from the patients.

ELIGIBILITY:
Inclusion criteria:

Subjects who will be recruited to this study are patients who met the criteria described below:

* Registered patients from September 2019 at Cipto Mangunkusumo Hospital
* Idiopathic uveitis patients (proven having negative result by available etiological uveitis work-ups) with IGRA positive. IGRA positive value is defined by score above 0.35 u/ml obtained from Quantiferon Tuberculosis (QFT)-Gold Assay (QIAGEN).
* Minimum age: 18 years old
* Proven not having active Tuberculosis
* Not previously received Anti Tuberculosis Therapy.
* Not consuming antibiotic one to two weeks prior to the time of study
* Not living together with Tuberculosis active patient
* Not having plan to become pregnant during the time of study
* Not part of reactive Tuberculosis risk group based on Latent Tuberculosis Incident WHO guidelines 2018
* Active inflammation in the past 180 days characterized by the following sign based on SUN Criteria(in at least one eye)

  * ≥ 2+ anterior chamber cells
  * ≥ 2+ vitreous haze
  * active retinal or choroidal lesions
* Active inflammation during patient registration, characterized by the following sign based on SUN Criteria (in at least one eye)

  * ≥1+ anterior chamber cells and/or
  * ≥1+ vitreous haze and/or
  * active retinal/choroidal lesions

Exclusion Criteria:

* Not willing to sign informed consent
* Pregnant patient
* Not coming to scheduled visit date
* Uveitis caused by infectious origin
* Media opacity caused by cataract and/ or corneal scar resulting in difficulty of posterior segment examination in both eyes
* Chronic hypotony (IOP < 5 mm Hg for > 3 months) in both eyes
* History of prior intraocular surgery in < 30 days, or arranged surgery within the next 6 months
* Best spectacle-corrected visual acuity (BSCVA) of hand motions or worse in better eye
* Any history of cancer excluding non-melanoma skin cancer
* Abnormal Complete blood count (≤ 2,500 white blood cells and/or ≤ 75,000 platelets and/or ≤9 hemoglobin) within 4 weeks prior to enrollment^
* Abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal for the lab and/or creatinine ≥ 1.5 within 4 weeks prior to enrollment^
* Patient with active infection of tuberculosis, HIV infection, syphilis, or hepatitis B or C

Note (^): Testing is conducted within 1-2 weeks prior to enrollment;

As many 10 subjects of the health volunteers are recruited for this study after giving consent. The health volunteers that will be recruited are the subject who met following criteria:

1. age: 18-50 years old (Man/Woman)
2. not having any health complaint or symptoms
3. not in any long term medication
4. body mass index: 18.5 - < 30
5. no history of allergy
6. willing to cooperate in this study
7. state of complete physical, mental, and social well being, and not merely the absence of disease or infirmity (WHO healthy definition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Idiopathic uveitis patients with IGRA positive registered from September 2019 at Cipto Mangunkusumo Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of clinical improvement | 0, 14 days, 8 weeks, 3 months, 6 months, and 12 months
  Clinical improvement of uveitis patients with IGRA positive after receiving complete Anti Tuberculosis Therapy is measured by using The Standardization of Uveitis Nomenclature (SUN) inflammation degree. Clinical improvement definition is decreasing of inflammation degree up to two degrees or becoming 0 degree. Meanwhile, clinical failure is defined by increasing of inflammation degree or decreasing of inflammation degree up to one degree/ not becoming 0 degree or unchanged degree of first to fourth degree.
The changes of type 1 interferon scoring in selected gene expression | 0, 14 days, 6 months.
  The score changes of type 1 interferon of uveitis patients with IGRA positive are determined by gene expression value of 10 varieties of type 1 interferon using Quantitative Reverse Transcriptase PCR (RT-qPCR) testing.

CONTACTS AND LOCATIONS:
Overall Officials: Rina La Distia Nora, Principal Investigator — Division of Ophthalmology Departement, Faculty of Medicine Universitas Indonesia
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta Pusat, Jakarta Special Capital Region, Indonesia